CLINICAL TRIAL: NCT00151983
Title: A Prospective, Open-Label, Multi-Center Study Evaluating the Safety and Tolerability of Methylphenidate Transdermal System (MTS) in Children Aged 6-12 Previously Treated With Extended-Release Methylphenidate Product.
Brief Title: Safety & Tolerability of MTS in Children Aged 6-12 Diagnosed With ADHD & Previously Treated With Extended-Release Methylphenidate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Collaborators: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD485-305
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate Transdermal System (Active Comparator): Methylphenidate 27.5mg, 41.3mg, 55mg, and 82.5mg patches applied daily for 8 weeks
  Interventions: Drug: Methylphenidate Transdermal System
- Placebo patch (Placebo Comparator): Placebo patch applied daily for 8 weeks
  Interventions: Drug: Methylphenidate Transdermal System

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — To assess the efficacy of 4- and 6-hour wear times of SPD485 (MTS) compared to placebo
  Other Names: MTS

SUMMARY:
This study will assess the safety and tolerability of MTS while attempting to establish the appropriate starting dose for subjects previously on an existing long-acting methylphenidate product.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a psychiatric disorder characterized by 3 main symptoms: inattention, hyperactivity and impulsivity. This study will assess the safety and tolerability of SPD485 while attempting to establish the appropriate starting dose for subjects previously on an existing long-acting methylphenidate product.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a primary diagnosis of ADHD
* Subject must be adequately controlled on a stable dose of one of the following medications for a 30 day period: Ritalin LA(r), Concerta(r), or Metadate DC(r), not to exceed 54 mg per day
* Females of childbearing potential must have a negative serum beta Human Chorionic Gonadotropin pregnancy test

Exclusion Criteria:

* A history of mental retardation that would indicate that the subject is not functioning at an age appropriate level intellectually
* A recent history of suspected substance abuse or dependence disorder
* Subject is taking Strattera
* Clinical signs and symptoms of skin irritation or hyper/hypopigmentation at the potential application sites

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2005-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Score on ADHD Rating Scale at 4 weeks | 30 days

SECONDARY OUTCOMES:
Parent rating scale | 30 days
Parent Global Assessment | 30 days
Medication Satisfaction Survey | 30 days
ADHD Impact Module | 30 days
Clinical Global Impressions Scale | 30 days
Adverse events, lab tests, dermal evaluations, ECGs | 30 days

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Meadowbrook Research, Inc., Scottsdale, Arizona
  - Psychiatric Centers at San Diego, San Marcos, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Miami Research Associates, Inc., Miami, Florida
  - Capstone Clinical Research, Libertyville, Illinois
  - Pedia Research, LLC, Owensboro, Kentucky
  - ProMed Pediatrics, Kalamazoo, Michigan
  - Children's Specialized Hospital, Toms River, New Jersey
  - North Carolina Neuropsychiatry PA, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations (OCCI, Inc.), Portland, Oregon
  - CNS Research Institute, Philadelphia, Pennsylvania
  - Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania
  - Claghorn-Lesem Research Clinic, Bellaire, Texas
  - ADHD Clinic of San Antonio, San Antonio, Texas
  - NeuroScience, Inc., Herndon, Virginia
  - Monarch Medical Research, Norfolk, Virginia

REFERENCES:
- [Derived] Bukstein OG, Arnold LE, Landgraf JM, Hodgkins P. Does switching from oral extended-release methylphenidate to the methylphenidate transdermal system affect health-related quality-of-life and medication satisfaction for children with attention-deficit/hyperactivity disorder? Child Adolesc Psychiatry Ment Health. 2009 Dec 10;3(1):39. doi: 10.1186/1753-2000-3-39. PMID 20003260
- [Derived] Arnold LE, Bozzolo DR, Hodgkins P, McKay M, Beckett-Thurman L, Greenbaum M, Bukstein O, Patel A. Switching from oral extended-release methylphenidate to the methylphenidate transdermal system: continued attention-deficit/hyperactivity disorder symptom control and tolerability after abrupt conversion. Curr Med Res Opin. 2010 Jan;26(1):129-37. doi: 10.1185/03007990903437412. PMID 19916704